CLINICAL TRIAL: NCT03894566
Title: NASCITA (Nascere E Crescere in Italia): an Italian Birth Cohort Study
Brief Title: NASCITA Italian Birth Cohort Study
Acronym: NASCITA
Status: Active, not recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: NASCITA; IRFMN 304 (Registry Identifier: Mario Negri Clinical Trials Registry)
Record Dates: First submitted 2019-03-12; First posted 2019-03-28 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Social Determinants of Health; Health Knowledge, Attitudes, Practice; Development, Child; Mental Disorders; Nutrition Disorders; Communicable Diseases
Keywords: Clinical Trial Protocol [Publication Type];; Cohort Studies; Infant, Newborn; Child; Infant; Health; Public Health; Predictors
MeSH Terms: conditions — Behavior; Mental Disorders; Nutrition Disorders; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention - birth cohort study — There are no interventions because it is a birth cohort study

SUMMARY:
The NASCITA study (NAscere e creSCere in ITAlia) was created to improve the understanding of the health status of Italian children early on and how it is affected by social and health determinants.

The study will evaluate physical, cognitive, and psychological development, and health status and health resource use during the first six years of life in a group of newborns, as well as potential associated factors. The association between the well-being of children and parental adherence to the recommendations for better child care and development will also be assessed.

Information on the children will be collected by paediatricians mostly during routine visits.

The findings will be used in the development of specific prevention measures and interventions to improve the health of children, in particular more vulnerable ones.

DETAILED DESCRIPTION:
The NASCITA study (NAscere e creSCere in ITAlia) was created to improve the understanding of the health status of Italian children early on and how it is affected by social and health determinants. The findings will be used in the development of specific prevention measures and interventions to improve the health of children, in particular more vulnerable ones.

The hypotheses are that:

* differences due to environmental, sociodemographic, and parental determinants, as well as to child characteristics and physician attitudes, exist between geographic areas in a population's health and in the use of health resources in the first few years of life;
* differences exist in the appropriateness of care provided by the National Health Service at different levels (regional, local, family pediatrician);
* differences exist between geographical settings in parental attitudes toward the recommendations concerning children's health care, and these differences may be a determinant of child development and well-being and health resource utilization;
* the existing differences between geographical settings in the opportunities for children to access educational/socialization experiences (e.g. day-care centers) may have an impact on development.

Aims:

* The main aim of the NASCITA cohort is to evaluate physical, cognitive, and psychological development, and health status and health resource use during the first six years of life in a group of newborns, and to evaluate potential associated factors.
* To evaluate differences between geographical settings in educational and socialization opportunities available for young children and in the care provided by the family pediatricians and by the National Health Service for the same needs
* To evaluate the association between the well-being of children and parental adherence to the recommendations for better child care and development.

More specifically:

* To evaluate child development through the monitoring of domains that affect nurturing care during the preschool period: health (disease prevention and treatment), nutrition (breastfeeding and dietary approach), safety and security (care and early intervention for vulnerable children), responsive caregiving (caregiving routine), and early learning (home opportunities to explore and learn);
* to identify potential factors influencing child well-being and growth and development, including the acquisition of competences.

The study population of the NASCITA cohort study will consist of children born in Italy during a one-year period who will be followed prospectively by participating pediatricians until at least the age of 6 years and whose parents agree to participate.

In Italy the large North-South divide is a major factor of socio-economic weakness and can be noted by the huge difference in statistical income between the northern and southern regions and municipalities.

Organization The coordination of the NASCITA study will be provided by the team of the Laboratory for Mother and Child Health of the Mario Negri Research Institute that integrates different expertise and competence with a long-standing experience in multicenter clinical research. The coordinating center will also carry out data collection, storage, management, and analysis. An independent scientific committee consisting of representatives of different disciplines and realities (including lay people) will monitor the development and results of the project.

NASCITA will be embedded in Italian pediatric primary care practice. A network of local contacts between pediatricians has been set up so that each node, representative of a setting, will act as a bridge to the coordinating center in conducting the study.

Recruitment The network that the study coordination center has built over the years involving hundreds of family pediatricians, documented by numerous collaborative publications, represents the first interlocutor to whom to propose participation in the study. The national Pediatric Cultural Association (ACP), with about 2000 members consisting mainly of family pediatricians, is among the supporters of the study. Pediatric scientific societies and associations will be contacted because detailed information concerning the study will be disseminated through national pediatric journals and internet-based resources. Recruitment will be based on the voluntary participation of interested pediatricians who can guarantee seven years of professional activity so that they can follow the enrolled newborns for the whole study period. This approach to enrolling pediatricians can be defined as a mixed method using also non-probability sampling techniques (convenience and purposive sampling) applied to choose a sample of subjects/units from a population.

Twenty-three geographic clusters were identified as representative of the country based on geographic and socio-economic characteristics and administrative divisions. Pediatricians and newborns of all the 23 identified clusters will be involved in the study.

Recruitment of the newborns (and their parents) will take place during the first routine well child visit scheduled for all newborns within their first 45 days of life at the office of the pediatrician assigned to them by the Local Health Units (LHU) to which they belong. Parents will receive oral and written information about the purpose and methods of the study and will be invited to participate.If they agree to participate, they will be asked to sign an informed consent. Recruitment of newborns will start in the first half of 2019, while recruitment of pediatricians will start in the preceding months.

Training and tutorial activities Before the start of the study, family pediatricians will be involved in training activities. Local coordinators will be trained by the research team, and will be responsible for the training of their peers at the local level. A CRF (case report form) was created in an online form with the contribution of local representatives of family pediatricians and scientific committee participants. During an initial phase, a group of family pediatricians tested the electronic CRF (eCRF), leading to improvements and adding the necessary questions to achieve an eCRF that would allow a more complete and simple collection of data. The eCRF will be available online before the start of the enrolment period in order to let participating family pediatricians familiarize with the information that needs to be collected.

Central and local monitoring of the study will be scheduled with the aim to guarantee follow up of the infants and the quality of data collected.

Data collection Data considered for the basic CRF are part of those routinely collected by the family pediatricians at the 7 standard well-child visits scheduled for all children during their first 6 years of life, and data collected during each contact with the enrolled children. However, expansion of the eCRF for specific research interests that may occur during the study period is foreseen. In order to enhance the quality of the data, the eCRF includes consistency and range checks to prevent internal inconsistencies, although the continuing review of collected data is guaranteed by the coordinating center and, in case of inconsistencies, pediatricians will be contacted. The administrators of the website (the coordinating center) will be able to view the completed forms also in a graphic format that will be updated periodically.

Baseline data At the first visit (within 45 days of life of the newborn), parents will be asked about parental medical history, characteristics and lifestyle, indoor and outdoor environment, and circumstances during pregnancy and around birth. Pregnancy and perinatal data will be collected also through hospital discharge documents following delivery.

Study population size The NASCITA cohort is sized to have enough power to study relatively common childhood exposures and outcomes, based on the national prevalence of certain health characteristics of Italian children and the expected number of cases for different enrolling scenarios. The aim is to recruit no less than 5000, and hopefully at least 10,000, newborns with complete information collected over the period of the study.

Analysis plan

In line with the aims of the study, univariate and multivariate analyses will be performed in an ongoing manner to investigate several associations in order to provide an answer to a number of research questions, including:

* the association between prenatal and living setting determinants and child neurocognitive development and health;
* the relationship between pregnancy, perinatal, and newborn growth characteristics and occurrence of adverse outcomes (i.e., obesity, hypertension, wheezing, eczema, hay fever, and asthma);
* the relationship between newborn and child nutrition quality and occurrence of overweight and obesity;
* the association between early stimulating learning initiatives and neurodevelopment of enrolled children;
* the association between vaccination and prevalence of preventable infectious diseases;
* the association between lifestyle factors and health inequalities and the trajectory of health in the preschool period.

Migrant newborns will be included in a special subgroup of analyses.

Materials produced A specific web portal for the NASCITA cohort study was developed (https://coortenascita.marionegri.it) to collect data, through a web-based form, and to provide findings and other information during the study period, also with the use of graphics on the analyses and data collected based on a successful approach already reported by the coordinating center.

Ethics and dissemination A consent form for participation will be signed by the pediatricians upon their first access to the web site. A paper consent form will be signed by parents at the first visit. This form includes the consent to data collection at each contact with the pediatrician during the six-year study period (first 6 years of the child's life). The filled in consent form will be stored by the pediatrician for ten years. Withdrawal from the study is guaranteed at any time both to pediatricians and parents. When consent is withdrawn, the child's data collected up to that point will be kept in the analyses, but no further data will be collected. Standard procedures for the protection of confidential individual information will be applied according to national and international ethical recommendations and guidelines as well as national legal regulations. Data will be pseudonymized and all analyses will be conducted with fully anonymized data sets.

A newsletter report will periodically be sent to the pediatricians and uploaded on the web site. During the study, different tools will be used to update the participating families mainly through the web site. Collected data will be periodically analyzed according to the aims of the project, and findings reported to lay people and the scientific community.

When the enrolled children reach the age of 6 years, if not decided otherwise in the meantime, their personal files will no longer be updated, but will be kept for another 10 years in the database.

NASCITA proposes to be a resource for the research community, so data will be available to public researchers outside the NASCITA research group upon request for collaborative research initiatives, after approval by the scientific committee.

ELIGIBILITY:
Inclusion Criteria:

* Family pediatricians who can guarantee seven years of professional activity
* Newborns seen by their family pediatrician for the first routine well-child visit within the first 45 days of life

Exclusion Criteria:

- Children not born in Italy

Max Age: 45 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Italian healthcare is provided through a network of Local Health Units, each of which consists of multiple healthcare districts. Every Italian resident is registered with a family (pediatric or general) practitioner. In Italy there are about 7500 family pediatricians, for an average of 450.000 births/year. About 60 newborns/year are therefore assigned to each pediatrician.
  Twenty-two geographic clusters were identified as representative of Italy based on geographic and socio-economic characteristics and administrative divisions. Pediatricians and newborns from all 22 clusters will be involved in the study. From the start of 2019, newborns will be continuously included in the study for an entire one-year period chosen by each pediatrician and will be followed until 6 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Height | Within 45 days of life
  Height in meters
Height | at 3 months of age
  Height in meters
Height | at 6 months of age
  Height in meters
Height | at 1 year of age
  Height in meters
Height | at 3 years of age
  Height in meters
Height | at 6 years of age
  Height in meters
Weight | Within 45 days of life
  Weight in kilograms
Weight | At 3 months of life
  Weight in kilograms
Weight | At 6 months of life
  Weight in kilograms
Weight | At 1 year of life
  Weight in kilograms
Weight | At 3 years of life
  Weight in kilograms
Weight | At 6 years of life
  Weight in kilograms
Child development | At 6 months of life
  Measured with the International Guide for Monitoring Child Development (GMCD), which involves 7 domains (language, fine and gross motor, relation, play and self-help) over 12 age periods from the 1st to the 42nd months. Each domain has specific age intervals that are met by typically developing children. If any of these are not met, a possible delay is noted. E.g. Fine motor (fine movements). "How does she use her hands and fingers, like holding objects?" [9-11 months]: Picks up small objects (like pieces of food using pincer (thumb and index finger) aided by other fingers. [12-14 months]: Picks up small objects using pincer (thumb and index finder) only.
Child development | At 1 year of life
  Measured with the International Guide for Monitoring Child Development (GMCD), which involves 7 domains (language, fine and gross motor, relation, play and self-help) over 12 age periods from the 1st to the 42nd months. Each domain has specific age intervals that are met by typically developing children. If any of these are not met, a possible delay is noted. E.g. Fine motor (fine movements). "How does she use her hands and fingers, like holding objects?" [9-11 months]: Picks up small objects (like pieces of food using pincer (thumb and index finger) aided by other fingers. [12-14 months]: Picks up small objects using pincer (thumb and index finder) only.
Child development | At 2 years of life
  Measured with the International Guide for Monitoring Child Development (GMCD), which involves 7 domains (language, fine and gross motor, relation, play and self-help) over 12 age periods from the 1st to the 42nd months. Each domain has specific age intervals that are met by typically developing children. If any of these are not met, a possible delay is noted. E.g. Fine motor (fine movements). "How does she use her hands and fingers, like holding objects?" [9-11 months]: Picks up small objects (like pieces of food using pincer (thumb and index finger) aided by other fingers. [12-14 months]: Picks up small objects using pincer (thumb and index finder) only.
Child development | At 3 years of life
  Measured with the International Guide for Monitoring Child Development (GMCD), which involves 7 domains (language, fine and gross motor, relation, play and self-help) over 12 age periods from the 1st to the 42nd months. Each domain has specific age intervals that are met by typically developing children. If any of these are not met, a possible delay is noted. E.g. Fine motor (fine movements). "How does she use her hands and fingers, like holding objects?" [9-11 months]: Picks up small objects (like pieces of food using pincer (thumb and index finger) aided by other fingers. [12-14 months]: Picks up small objects using pincer (thumb and index finder) only.
Child development | At 6 years of life
  Measured with the International Guide for Monitoring Child Development (GMCD), which involves 7 domains (language, fine and gross motor, relation, play and self-help) over 12 age periods from the 1st to the 42nd months. Each domain has specific age intervals that are met by typically developing children. If any of these are not met, a possible delay is noted. E.g. Fine motor (fine movements). "How does she use her hands and fingers, like holding objects?" [9-11 months]: Picks up small objects (like pieces of food using pincer (thumb and index finger) aided by other fingers. [12-14 months]: Picks up small objects using pincer (thumb and index finder) only.
Incidence of child overweight and obesity | At 3 years of life
  Measured as BMI in kg/m^2
Incidence of child overweight and obesity | At 6 years of life
  Measured as BMI in kg/m^2
Duration of exclusive breastfeeding | Within 45 days of life
  The paediatrician will ask the mother if she is still exclusively breastfeeding
Duration of exclusive breastfeeding | At 3 months of life
  The paediatrician will ask the mother if she is still exclusively breastfeeding
Duration of exclusive breastfeeding | At 6 months of life
  The paediatrician will ask the mother if she is still exclusively breastfeeding
Number of children with wheezing episodes | At 2 years of life
  Number of children who have had at least one wheezing episode
Number of children with wheezing episodes | At 3 years of life
  Number of children who have had at least one wheezing episode
Number of children with asthma | At 6 years of life
  Number of children who have asthma
Number of respiratory tract infection episodes in the preschool period | At 1 year of life
  Number of respiratory tract infection episodes
Number of respiratory tract infection episodes in the preschool period | At 2 years of life
  Number of respiratory tract infection episodes
Number of respiratory tract infection episodes in the preschool period | At 3 years of life
  Number of respiratory tract infection episodes
Number of respiratory tract infection episodes in the preschool period | At 6 years of life
  Number of respiratory tract infection episodes
Number of hospitalizations | At 1 year of life
  The paediatrician will ask the mother about the number of hospitalizations
Number of hospitalizations | At 2 years of life
  The paediatrician will ask the mother about the number of hospitalizations
Number of hospitalizations | At 6 years of life
  The paediatrician will ask the mother about the number of hospitalizations
Childhood vaccinations | At 3 months of life
  The paediatrician will note which vaccines the child has received so far
Childhood vaccinations | At 6 months of life
  The paediatrician will note which vaccines the child has received so far
Childhood vaccinations | At 1 year of life
  The paediatrician will note which vaccines the child has received so far
Childhood vaccinations | At 2 years of life
  The paediatrician will note which vaccines the child has received so far
Childhood vaccinations | At 6 years of life
  The paediatrician will note which vaccines the child has received so far
Maternal vaccinations in pregnancy | Within 45 days of life of the child
  The paediatrician will ask the mothers which vaccines they received during the pregnancy

SECONDARY OUTCOMES:
Hearing test | At 6 months of life
  Assessed with the Boel test

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Bonati, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri; Antonio Clavenna, MD, PhD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri; Chiara Pandolfini, BA, PhD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Istituto di Ricerche Farmacologiche Mario Negri IRCCS, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
The scientific committee will evaluate single requests for data

REFERENCES:
- [Background] Pandolfini C, Clavenna A, Campi R, Cartabia M, Finazzi S, Bonati M. Parental practices that influence children's development: how often are they implemented and by whom-results from the NASCITA birth cohort study. Eur J Pediatr. 2024 Jul;183(7):3029-3038. doi: 10.1007/s00431-024-05564-w. Epub 2024 Apr 22. PMID 38644455
- [Background] Pansieri C, Clavenna A, Pandolfini C, Zanetti M, Calati MG, Miglio D, Cartabia M, Zanetto F, Bonati M. NASCITA Italian birth cohort study: a study protocol. BMC Pediatr. 2020 Feb 19;20(1):80. doi: 10.1186/s12887-020-1961-1. PMID 32075601
- [Background] Zanetti M, Clavenna A, Pandolfini C, Pansieri C, Calati MG, Cartabia M, Miglio D, Bonati M. Informatics Methodology Used in the Web-Based Portal of the NASCITA Cohort Study: Development and Implementation Study. J Med Internet Res. 2021 Mar 12;23(3):e23087. doi: 10.2196/23087. PMID 33709930
- [Background] Pandolfini C, Clavenna A, Cartabia M, Campi R, Bonati M; NASCITA Work Group. National, longitudinal NASCITA birth cohort study to investigate the health of Italian children and potential influencing factors. BMJ Open. 2022 Nov 15;12(11):e063394. doi: 10.1136/bmjopen-2022-063394. PMID 36379649
- [Background] Clavenna A, Morabito E, Cartabia M, Campi R, Pandolfini CL, Bonati M; NASCITA Working Group. National, longitudinal NASCITA birth cohort study: prevalence of overweight at 12 months of age in children born healthy. BMJ Paediatr Open. 2023 Jan;7(1):e001622. doi: 10.1136/bmjpo-2022-001622. PMID 36625429
- [Derived] Segre G, Clavenna A, Cartabia M, Bonati M; NASCITA Working Group. Postpartum depression screening in mothers and fathers at well-child visits: a feasibility study within the NASCITA cohort. BMJ Open. 2023 Jun 23;13(6):e069797. doi: 10.1136/bmjopen-2022-069797. PMID 37355274
- See also: NASCITA Cohort website — https://nascita.marionegri.it/